CLINICAL TRIAL: NCT02062138
Title: Effectiveness of New Interventional Approaches to Improve Physical Function Following Total Knee Arthroplasty
Brief Title: Effectiveness of Passive and Active ROM Exercises Following TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Anett Mau-Moeller, M.A., University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPAB
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty
Keywords: rehabilitation; total knee arthroplasty; range of motion; continuous passive motion; controlled active motion; postoperative physical therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- continuous passive motion (CPM) (Active Comparator)
  Interventions: Other: continuous passive motion (CPM)
- controlled active motion (CAM I) (Experimental)
  Interventions: Other: controlled active motion (CAM I)
- controlled active motion (CAM II) (Experimental)
  Interventions: Other: controlled active motion (CAM II)

INTERVENTIONS:
Other: continuous passive motion (CPM) — standard-of-care therapy (control intervention); Patients receive three 30 minutes CPM applications (unilateral op-leg) each day from the second postoperative day until 1 day prior to discharge.
  Arms: continuous passive motion (CPM)
Other: controlled active motion (CAM I) — Patients receive three 30 minutes CAM applications (unilateral op-leg) each day from the second postoperative day until 1 day prior to discharge.
  Arms: controlled active motion (CAM I)
Other: controlled active motion (CAM II) — Patients receive three 30 minutes CAM applications (bilateral alternating) each day from the second postoperative day until 1 day prior to discharge.
  Arms: controlled active motion (CAM II)

SUMMARY:
The purpose of the study is to determine the effectiveness of new interventional approaches in the early postoperative phase following total knee arthroplasty (TKA). It is assumed that active training programs are more effective in improving physical function than the passive standard-of-care therapy.

DETAILED DESCRIPTION:
The major objectives of rehabilitation after TKA are the early regain of range of motion (ROM) and mobilization of the patient. Continuous passive motion (CPM) is frequently used as part of the postoperative care regime following TKA with the aim to increase knee joint mobility and improve postoperative recovery despite little conclusive scientific evidence. Conflicting research findings have generated an ongoing debate on its usage. As the greatest loss of function occurs in the first month following TKA, it is surprising that the ROM therapy during hospital stay is still carried out passively. A passive mobilization of the knee joint with CPM does not encourage the patients to actively participate in their rehabilitation. Research on the effectiveness of active ROM exercises added to standard physiotherapy during the short in-hospital period is lacking so far.The objective of this study is to compare the passive clinical standard therapy (CPM) with different active training programs (controlled active motion, CAM). It was hypothesised that the CAM therapies are more effective in improving physical function than the CPM therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis and scheduled for primary TKA
* age: 50-80

Exclusion Criteria:

* BMI > 40
* musculoskeletal and neurological disorders that limit physical function
* any planned further joint surgery within 6 months
* substantial pain or functional limitation which make the patients unable to perform study procedures

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
range of motion | change from baseline (before surgery) to discharge (9 days post surgery)

SECONDARY OUTCOMES:
neuromuscular function | change from baseline (before surgery) to discharge (9 days after surgery)
joint position sense | change from baseline (before surgery) to discharge (9 days after surgery)
motor function | change from baseline (before surgery) to discharge (9 days after surgery)
  stair climbing test, timed up and go test
cognitive functioning | change from baseline (before surgery) to discharge (9 days after surgery)
physical activity | change from baseline (before surgery) to discharge (9 days after surgery)
  over a period of 7 days using the activPAL activity recording system.
pain | change from baseline (before surgery) to discharge (9 days after surgery)
  visual analogue scale (VAS)
swelling | change from baseline (before surgery) to discharge (9 days after surgery)
length of hospital stay | change from baseline (before surgery) to discharge (9 days after surgery)
quality of life | change from baseline (before surgery) to discharge (9 days after surgery)
  36-item Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Bader, MD, Study Chair — Department of Orthopedics, University Medicine Rostock; Ralf Skripitz, MD, Study Director — Department of Orthopedics, University Medicine Rostock; Anett Mau-Moeller, M.A., Principal Investigator — Department of Orthopedics, University Medicine Rostock; Martin Behrens, Principal Investigator — Department of Kinesiology, University of Rostock; Tino Stöckel, PhD, Principal Investigator — Department of Kinesiology, University of Rostock
Locations (1):
- Department of Orthopedics, University Medicine Rostock, Rostock, Germany

REFERENCES:
- [Derived] Jacksteit R, Stockel T, Behrens M, Feldhege F, Bergschmidt P, Bader R, Mittelmeier W, Skripitz R, Mau-Moeller A. Low-Load Unilateral and Bilateral Resistance Training to Restore Lower Limb Function in the Early Rehabilitation After Total Knee Arthroplasty: A Randomized Active-Controlled Clinical Trial. Front Med (Lausanne). 2021 Jun 22;8:628021. doi: 10.3389/fmed.2021.628021. eCollection 2021. PMID 34239883